CLINICAL TRIAL: NCT02913989
Title: Characterization of Smoking Habits Patterns in Medical Doctors of a Central Hospital in Portugal - What Has Changed After 15 Years? A Comparative Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar Lisboa Ocidental (Other Government)
Responsible Party: Principal Investigator, Rafaela Campanha, MD, Centro Hospitalar Lisboa Ocidental
Other Study IDs: 1
Record Dates: First submitted 2016-09-13; First posted 2016-09-26 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Smoking Cessation; Tobacco Dependence
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Doctors from Medical Specialities: Doctors from Medical Specialities A voluntary and anonymous questionnaire was distributed to all physicians for a period of 4 months. The questions included sociodemographic data, smoking habits characterization, attitudes towards smoking, importance attribute to smoking cessation programme in the hospital and knowledge of the 2008 country law.
  Interventions: Other: Smoking habits characterization
- Doctors from Surgical Specialities: Doctors from Surgical Specialities A voluntary and anonymous questionnaire was distributed to all physicians for a period of 4 months. The questions included sociodemographic data, smoking habits characterization, attitudes towards smoking, importance attribute to smoking cessation programme in the hospital and knowledge of the 2008 country law.
  Interventions: Other: Smoking habits characterization

INTERVENTIONS:
Other: Smoking habits characterization

SUMMARY:
Abstract: Tobacco dependence remains one of the primary health care concerns worldwide. Attitude of healthcare professionals towards smoking is crucial for any long-term prevention and smoking cessation program.

Objectives: Analyze smoking habits of medical doctors from a central hospital in Lisbon (2014), comparing results between medical versus surgical specialities. Results were compared with those obtained in 1999.

Design and setting: A voluntary and anonymous questionnaire was distributed to all physicians for a period of 4 months. The questions included sociodemographic data, smoking habits characterization, attitudes towards smoking, importance attribute to smoking cessation programme in the hospital and knowledge of the 2008 country law.

Participants: All medical doctors working in the central hospital studied between 1/1/2014 and 30/6/2014 Outcome measures: The primary outcome measure was to characterize the smoking habits of medical doctors. Secondary outcomes included comparison of results between surgical and medical groups and with those obtain in a similar study in 1999.

ELIGIBILITY:
Inclusion Criteria:

* All medical doctors working in the central hospital studied between 1/1/2014 and 30/6/2014

Exclusion Criteria:

* Not a medical doctor

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All medical doctors working in the central hospital studied between 1/1/2014 and 30/6/2014
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Analyze smoking habits of medical doctors from a central hospital in Lisbon (2014), comparing results between medical versus surgical specialities. | 1 March 2014 - 30 June 2014

SECONDARY OUTCOMES:
Comparison of smoking habits of medical doctors in 2014 with a similar study in 1999 in the same hospital. | 1999 and 2014 - 15 years